CLINICAL TRIAL: NCT05847413
Title: Targeting Beta Cell Dysfunction With Verapamil in Longstanding T1D
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB20042
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Verapamil

STUDY DESIGN:
Intervention Model Description: open label proof of concept study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Targeting Beta cell Dysfunction with Verapamil in Longstanding T1D (Experimental): Participants will receive verapamil for 12 weeks
  Interventions: Drug: Verapamil

INTERVENTIONS:
Drug: Verapamil — Subjects will receive oral verapamil for 12 weeks

SUMMARY:
The purpose of this study is to determine whether verapamil can transiently improve beta cell function in those who do or do not secrete proinsulin and little/no C-peptide.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 3 years from Type 1 diabetes diagnosis
2. Males and females 18-50 years of age, inclusive
3. Peak MMTT stimulated C-peptide < 0.017 pmol/mL
4. Females of child-bearing potential must be willing to use effective birth control for 12 weeks
5. Willing and able to give informed consent for participation
6. HbA1c ≤ 8.5%

Exclusion Criteria:

* Concurrent use of non-insulin therapies aimed to control hyperglycemia or use within the past 30 days of initial qualifying MMTT (V-2). 2. Diagnosis of liver disease or elevated hepatic enzymes, as defined by ALT or AST> 1.5 x the upper limit of age-determined normal (ULN). 3. Renal disease, as defined by creatinine ≥1.5 mg/dL. 4. Hypersensitivity to verapamil or any component of the formulation. 5. Previous use of verapamil. 6. Known left ventricular dysfunction; bradycardia (HR <50 BPM) hypotension (systolic pressure <90 mm Hg); PR interval prolongation on EKG or any bradyarrhythmia (e.g. sick sinus syndrome, Anterior Ventral (AV) block); atrial flutter or fibrillation, and an accessory bypass tract (Wolff- Parkinson- White (WPW) syndrome, Lown-Ganong-Levine syndrome) 7. Uncompensated heart failure, fluid overload, myocardial infarction or evidence of ischemic heart disease or other serious cardiac disease as described in New York Heart Association (NYHA) Class III or IV criteria within the 12 weeks before randomization. 8. Use of beta blockers or medium-high dose statins: any dose of atorvastatin (Lipitor) or rosuvastatin (Crestor); simvastatin > 10 mg daily; lovastatin > 20 mg; pravastatin > 20 mg 9. Use of other medications which may increase the concurrent risk of verapamil use, including medications which utilize the cytochrome p450 enzyme pathway. 10. Females who are pregnant or lactating. 11. Receipt of an immune modulating biologic or investigational drug within 3 months or 5 half-lives before enrollment. 12. History of other clinically significant autoimmune disease except for celiac and stable thyroid disease. 13. Current use of any medication known to significantly influence glucose tolerance (e.g. oral steroids, atypical antipsychotics, diphenylhydantoin, niacin). 14. Any medical or psychological condition that in the opinion of the principal investigator would interfere with the safe completion of the trial. Conditions to consider include history of chronic GERD, chronic constipation, and chronic nausea. 15. Specific to MRI subjects: non-removable ferromagnetic materials or MRI not technically feasible (claustrophobia, movement disorder, obesity).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Proportion of individuals with peak MMTT stimulated C-peptide >0.017 pmol/mL at 12 weeks. | 0-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carla Greenbaum, MD, Principal Investigator — Benaroya Research Institute
Locations (1):
- Benaroya Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lord SM, Bahnson HT, Greenbaum CJ, Liljenquist DR, Virostko J, Speake C. Testing a new platform to screen disease-modifying therapy in type 1 diabetes. PLoS One. 2023 Dec 14;18(12):e0293268. doi: 10.1371/journal.pone.0293268. eCollection 2023. PMID 38096190